CLINICAL TRIAL: NCT06743945
Title: A Prospective, Multicenter, Phase II Study of POLA-R-CHP in the First-line Treatment of Transformed DLBCL
Brief Title: POLA-R-CHP in the First-line Treatment of Transformed DLBCL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Yizhen Liu, Clinical Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: iNHL-05
Record Dates: First submitted 2024-12-15; First posted 2024-12-20 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Transformed Lymphoma
MeSH Terms: interventions — polatuzumab vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): POLA-R-CHP
  Interventions: Drug: POLA-R-CHP

INTERVENTIONS:
Drug: POLA-R-CHP — Pola-R-CHP is a combination of rituximab, cyclophosphamide, doxorubicin, prednisone, and polatuzumab vedotin
  Other Names: polatuzumab vedotin and R-CHP

SUMMARY:
This study aims to evaluate efficacy and safety of POLA-R-CHP in the treatment of patients with transformed DLBCL.

DETAILED DESCRIPTION:
Patients with transformed DLBCL lack standard treatment. We intend to conduct a prospective, multicenter, phase II study in order to evaluate efficacy and safety of POLA-R-CHP as first-line treatment of patients with transformed DLBCL.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 -80 years old;
* Histologically confirmed transformed DLBCL;
* ECOG 0-2;
* Signed informed consent form.
* Having sufficient organ function: a) Hematopoietic function: Neutrophils ≥ 1.0 × 109/L, PLT ≥ 75 × 109/L, Hb ≥ 90g/L(unless caused by underlying disease, as judged by the investigator, such as extensive bone marrow involvement, or hypersplenism secondary to lymphoma splenic involvement); b) Liver function: bilirubin ≤1.5 times the upper limit of normal (ULN), ALT and AST<3 x ULN, serum albumin ≥ 30 g/L; c) Renal function: serum Cr<1.5 × ULN, creatinine clearance rate ≥ 50mL/min (calculated according to the standard Cockcroft Gault formula, if renal dysfunction is caused by tumor compression, creatinine clearance rate ≥ 30mL/min); d) Left ventricular ejection fraction (LVEF) ≥ 50% detected by echocardiography.

Exclusion Criteria:

* Individuals who are allergic to human or mouse monoclonal antibodies, or known sensitivity or allergic reaction to murine products;
* Previous organ transplantation;
* Prior treatment of any condition (e.g., cancer, rheumatoid arthritis) with cytotoxic drugs within 5 years at the time of screening or prior use of any anti-CD20 antibodies;
* Evidence of uncontrolled significant comorbidities that may affect the patient's compliance with the study protocol or affect the interpretation of the study results, including significant cardiovascular disease (such as New York College of Cardiology Class III or IV heart disease, myocardial infarction within the past 6 months, unstable arrhythmia, or unstable angina) or pulmonary disease (including history of obstructive pulmonary disease and bronchospasm);
* Recent major surgery (within 4 weeks prior to enrollment), excluding diagnostic surgery;
* Known active bacterial, viral, fungal, mycobacterial, parasitic or other infections (except for fungal infections in nail beds) at the time of study enrollment or major infections within 2 weeks before the start of the first course of treatment;
* Previous radiotherapy in the mediastinum/pericardial region;
* Active chronic hepatitis B infection (defined as HBV DNA positive): If hepatitis B virus (HBV) DNA cannot be detected during screening, patients with latent or previous hepatitis B infection (defined as positive hepatitis B surface antigen or hepatitis B core total antibody) can be included in this study. The above patients must voluntarily undergo regular HBV-DNA testing and receive appropriate antiviral treatment according to regulations.
* For patients with positive hepatitis C virus (HCV) antibody serological test, only when polymerase chain reaction (PCR) shows negative HCV-RNA can participate in this study.
* Patients with active HIV and syphilis infections;
* Pregnant or lactating women;
* The researcher determined that patients are not suitable to participate in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
2-year progression-free survival (PFS) assessed by imaging examination | From date of patients sign informed consent until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  the period from the date of patients sign informed consent to the observed progression of the disease or the occurrence of death for any reason

SECONDARY OUTCOMES:
complete remission rate assessed by imaging examination | up to 6 months
  the ratio of numbers of patients with complete response after 6 treatment cycles to all the participants
2-year event-free survival (EFS) | From date of patients sign informed consent until the date of first documented event, progression or date of death from any cause, whichever came first, assessed up to 2 years
  the period from the date of patients sign informed consent to the observed event for any reason
2-year overall survival rate | From date of patients sign informed consent until the date of death or the date of last follow-up time, whichever came first, assessed up to 2 years
  time between the date of patients sign informed consent and the date of death or the date of last follow-up time
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Through study completion, up to 2 years
  number of participants with treatment-related adverse events as assessed by CTCAE v5.0

OTHER OUTCOMES:
tissue biomarkers | Throughout the treatment period, up to 2 years
  Detection of tissue DNA biomarkers in the treatment of transformed diffuse large B cell lymphoma

CONTACTS AND LOCATIONS:
Overall Officials: Yizhen Liu, M.D., Ph.D., Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No